CLINICAL TRIAL: NCT04260815
Title: The Effect of Transcranial Direct-current Stimulation on Discourse Production in Healthy Older Adults
Brief Title: The Effect of Non-invasive Brian Stimulation on Language Production in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HR-19/20-6391
Record Dates: First submitted 2020-01-29; First posted 2020-02-07 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Language Disorders; Aphasia; Stroke
MeSH Terms: conditions — Language Disorders; Aphasia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anodal tDCS on the left inferior frontal gyrus (IFG) (Experimental)
  Interventions: Device: Transcranial direct-current stimulation (tDCS)
- anodal tDCS on the right IFG (Experimental)
  Interventions: Device: Transcranial direct-current stimulation (tDCS)
- sham tDCS (Sham Comparator)
  Interventions: Device: Transcranial direct-current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct-current stimulation (tDCS) — Transcranial direct-current stimulation is a non-invasive brain stimulation method that can modify spontaneous cortical activity in targeted brain regions. Anodal tDCS delivered through a positively charged electrode has been found to increase cortical excitability in a targeted brain region. Application of tDCS has been found to improve language production in healthy and brain-injured speakers.

SUMMARY:
The use of non-invasive brain stimulation techniques like transcranial direct-current stimulation (tDCS) for rehabilitation of language is a growing field that needs further studies to determine how best it can be used to enhance treatment outcomes. It has been shown that tDCS can improve language performance in healthy and brain-injured individuals such as increased naming accuracy.

However, at present, it is not known what effect tDCS has on higher-level language skills like discourse production (i.e. story telling, giving instructions) in healthy, older speakers. Therefore, the aim of this study is to investigate in healthy older adults, the effect of tDCS on discourse production as well as the ideal tDCS electrode placement for improving language at the discourse level. It is hypothesised that tDCS will result in greater language changes and improvements during discourse production compared to no stimulation.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years of age
* Native English speakers
* Right handed
* Normal aided or unaided visual acuity
* At least secondary school level of education

Exclusion Criteria:

* History of neurological disease or cognitive impairment
* Any contraindication of tDCS (i.e. history of seizures, metal implants)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Change in word total | pre-intervention and immediately after the intervention
  total number of words in a language sample
Change in verb total | pre-intervention and immediately after the intervention
  total number of verbs in a language sample
Change in utterance total | pre-intervention and immediately after the intervention
  total number of utterances (complete sentences including a predicate and argument) in a language sample
Change in percent of Correct Information Units | pre-intervention and immediately after the intervention
  The percent of accurately produced words that provide information relevant to the language task

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 7 days
  HADS is a 14-item scale which assesses non-somatic anxiety and depression symptoms experienced in the past week. Scores range from 0 to 21 for each sub-scale with a score ≥8 proposed for the identification of caseness, for both depression and anxiety.
EPIC Physical Activity Questionnaire (EPAQ2) | 12 months
  The EPAQ2 is a self completed questionnaire which collects information on a person's physical activity levels at home, work and recreation. Based on total activity hours in the last 12 months, the physical activity index categorises levels of physical activity into 'active', 'moderately inactive', 'moderately active' or 'active'.
The Keele Assessment of Participation (KAP) | 4 weeks
  The KAP is a short questionnaire that measures participation levels in various activities such as activities of daily living, social activities and work in the last 4 weeks. A score of 0 indicates no restriction in participation whereas scores from 1-11 indicate a restriction in participation in at least one activity ( the higher the score the greater the restriction).

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All information collected will be kept confidential and stored anonymously on password protected computers used only by research staff who are part of the study. Data will be stored securely in accordance with the Data Protection Act (1998) and the General Data Protection Regulations (May 2018). Stored, anonymised data may be used for future medical and health-related studies. Anonymised data will be retained for 10 years.

REFERENCES:
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Thair H, Holloway AL, Newport R, Smith AD. Transcranial Direct Current Stimulation (tDCS): A Beginner's Guide for Design and Implementation. Front Neurosci. 2017 Nov 22;11:641. doi: 10.3389/fnins.2017.00641. eCollection 2017. PMID 29213226
- [Background] Cattaneo Z, Pisoni A, Papagno C. Transcranial direct current stimulation over Broca's region improves phonemic and semantic fluency in healthy individuals. Neuroscience. 2011 Jun 2;183:64-70. doi: 10.1016/j.neuroscience.2011.03.058. Epub 2011 Apr 6. PMID 21477637
- [Background] Saffran EM, Berndt RS, Schwartz MF. The quantitative analysis of agrammatic production: procedure and data. Brain Lang. 1989 Oct;37(3):440-79. doi: 10.1016/0093-934x(89)90030-8. PMID 2804622
- [Background] Monti A, Ferrucci R, Fumagalli M, Mameli F, Cogiamanian F, Ardolino G, Priori A. Transcranial direct current stimulation (tDCS) and language. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):832-42. doi: 10.1136/jnnp-2012-302825. Epub 2012 Nov 8. PMID 23138766
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Wilkie R, Peat G, Thomas E, Hooper H, Croft PR. The Keele Assessment of Participation: a new instrument to measure participation restriction in population studies. Combined qualitative and quantitative examination of its psychometric properties. Qual Life Res. 2005 Oct;14(8):1889-99. doi: 10.1007/s11136-005-4325-2. PMID 16155776
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Wareham NJ, Jakes RW, Rennie KL, Mitchell J, Hennings S, Day NE. Validity and repeatability of the EPIC-Norfolk Physical Activity Questionnaire. Int J Epidemiol. 2002 Feb;31(1):168-74. doi: 10.1093/ije/31.1.168. PMID 11914316